CLINICAL TRIAL: NCT00943761
Title: A Phase II Open Label Study of MK-7009 Administered Concomitantly With Pegylated Interferon Alfa-2a and Ribavirin to Patients With Chronic Hepatitis C Infection After Participation in Other MK-7009 Clinical Trials
Brief Title: A Study of Vaniprevir (MK-7009) in Participants With Chronic Hepatitis C Infection After Participation in Other Vaniprevir Studies (MK-7009-028)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7009-028; 2009_615 (Other: Merck); 2009-013053-15 (EudraCT Number)
Record Dates: First submitted 2009-07-21; First posted 2009-07-22 (Estimated); Results first posted 2014-09-29 (Estimated); Last update posted 2021-02-08 (Actual); Status verified 2021-01

CONDITIONS: Hepatitis C, Chronic
Keywords: hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — vaniprevir; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vaniprevir 300 mg b.i.d. + peg-IFN + RBV (Experimental): Participants received vaniprevir 300 mg twice daily (b.i.d.) in combination peg-IFN 180 mcg weekly and ribavirin (1000 or 1200 mg) administered as a divided dose twice daily.
  Interventions: Drug: Vaniprevir 300 mg b.i.d.; Drug: Pegylated interferon; Drug: Ribavirin
- Vaniprevir 600 mg b.i.d. + peg-IFN + RBV (Experimental): Participants received vaniprevir 600 mg b.i.d. in combination peg-IFN 180 mcg weekly and ribavirin (1000 or 1200 mg) administered as a divided dose twice daily.
  Interventions: Drug: Vaniprevir 600 mg b.i.d.; Drug: Pegylated interferon; Drug: Ribavirin

INTERVENTIONS:
Drug: Vaniprevir 600 mg b.i.d. — Oral capsules containing 150 mg vaniprevir, four in the morning and four in the evening, for 48 weeks
  Arms: Vaniprevir 600 mg b.i.d. + peg-IFN + RBV
Drug: Vaniprevir 300 mg b.i.d. — Oral capsules containing 150 mg vaniprevir, two in the morning and two in the evening, for 48 weeks
  Arms: Vaniprevir 300 mg b.i.d. + peg-IFN + RBV
Drug: Pegylated interferon — Prefilled syringe containing 180 µg/0.5 mL peg-IFN, for weekly subcutaneous injection, for 48 weeks
  Other Names: PEGASYS™
Drug: Ribavirin — Oral tablets containing 200 mg RBV, 5 or 6 tablets, dosage based on the participant's weight (<75 kg or ≥75 kg, respectively), for 48 weeks
  Other Names: COPEGUS™

SUMMARY:
This study will provide vaniprevir 600 mg or 300 mg twice daily in combination with pegylated interferon (peg-IFN) and ribavirin (RBV) to participants with chronic hepatitis C virus (HCV) infection who did not achieve viral eradication while participating in a prior vaniprevir clinical trial (MK-7009-004, NCT00518622; MK-7009-007, NCT00704405; MK-7009-009, NCT00704184; and MK-7009-029, NCT00954993).

ELIGIBILITY:
Inclusion criteria:

* Participant has participated in a prior vaniprevir clinical trial
* Participant agrees to use acceptable birth control method during treatment

Exclusion criteria:

* More than one year has passed since the participant was determined to be eligible for enrollment in protocol 028
* Participant discontinued vaniprevir and/or peg-IFN and/or RBV in the prior study due to a safety or tolerability issue
* Participant received any investigational therapy for HCV after participating in the prior study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2009-10-23 (Actual); Primary Completion 2013-05-29 (Actual); Study Completion 2013-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=7009-028&kw=7009-028&tab=access

RESULTS

PARTICIPANT FLOW:
Groups:
- Vaniprevir 300 mg b.i.d. + Peg-IFN + RBV: Participants received vaniprevir 300 mg twice daily in combination pegylated interferon (peg-IFN) 180 mcg weekly and ribavirin (RBV) 1000 or 1200 mg administered as a divided dose twice daily.
- Vaniprevir 600 mg b.i.d. + Peg-IFN + RBV: Participants received vaniprevir 600 mg twice daily in combination peg-IFN 180 mcg weekly and ribavirin 1000 or 1200 mg administered as a divided dose twice daily.
Period: Overall Study
Arm/Group | Vaniprevir 300 mg b.i.d. + Peg-IFN + RBV | Vaniprevir 600 mg b.i.d. + Peg-IFN + RBV
Started | 21 | 24
Completed | 17 | 23
Not Completed | 4 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Vaniprevir 300 mg b.i.d. + Peg-IFN + RBV: Participants received vaniprevir 300 mg twice daily in combination peg-IFN 180 mcg weekly and RBV 1000 or 1200 mg administered as a divided dose twice daily.
- Total: Total of all reporting groups
Arm/Group | Vaniprevir 300 mg b.i.d. + Peg-IFN + RBV | Vaniprevir 600 mg b.i.d. + Peg-IFN + RBV | Total
Number analyzed (Participants) | 21 | 24 | 45
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.5 (7.4) | 48.1 (8.4) | 50.2 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 14 | 20 | 34

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced an Adverse Event
Description: An adverse event is any unfavorable and unintended change in the structure, function, or chemistry of the body whether or not considered related to the study treatment.
Time Frame: up to 72 weeks
Population: All participants as treated population consists of all participants who received at least one dose of study treatment.
Measure: Number; unit: Participants
Arm/Group | Vaniprevir 300 mg b.i.d. + Peg-IFN + RBV | Vaniprevir 600 mg b.i.d. + Peg-IFN + RBV
Number analyzed (Participants) | 21 | 24
Participants | 21 | 23

2. Primary Outcome: Number of Participants Who Experienced a Serious Adverse Event
Description: Serious adverse event is defined as any adverse drug or biologic or device experience occurring at any dose resulting in death, was life-threatening, was persistent or caused significant disability/incapacity, required in-patient hospitalization or prolonged hospitalization, was a congenital anomaly or birth defect, was a cancer, or was an overdose.
Time Frame: up to 72 weeks
Population: All participants as treated population consists of all participants who received at least one dose of study treatment.
Measure: Number; unit: Participants
Arm/Group | Vaniprevir 300 mg b.i.d. + Peg-IFN + RBV | Vaniprevir 600 mg b.i.d. + Peg-IFN + RBV
Number analyzed (Participants) | 21 | 24
Participants | 4 | 1

3. Primary Outcome: Number of Participants Who Discontinued Study Treatment Due to an Adverse Event
Description: as for outcome 1
Time Frame: 48 weeks
Population: All participants as treated population consists of all participants who received at least one dose of study treatment.
Measure: Number; unit: Participants
Arm/Group | Vaniprevir 300 mg b.i.d. + Peg-IFN + RBV | Vaniprevir 600 mg b.i.d. + Peg-IFN + RBV
Number analyzed (Participants) | 21 | 24
Participants | 2 | 1

4. Primary Outcome: Percentage of Participants Who Achieved Sustained Viral Response 24 Weeks After the End of Treatment (SVR24)
Description: SVR24 is defined as undetectable hepatitis C virus ribonucleic acid (HCV RNA) 24 weeks after the end of vaniprevir study therapy. HCV RNA plasma levels were assessed using the Roche COBAS Taqman assay (or equivalent) with the limit of quantification (LoQ) of at least 25 IU/mL and the limit of detection (LoD) of at least 10 IU/mL.
Time Frame: 72 weeks
Population: Population includes only a subset of participants previously treated with placebo + peg-IFN + RBV in a vaniprevir study and excludes participants for failure to receive >=1 dose of study drug, lack of any post-allocation endpoint data subsequent to >=1 dose of study drug, lack of baseline data, or missing data due to discontinuation from the study
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Vaniprevir 300 mg b.i.d. + Peg-IFN + RBV | Vaniprevir 600 mg b.i.d. + Peg-IFN + RBV
Number analyzed (Participants) | 18 | 17
Percentage of participants | 66.7 [41.0 to 86.7] | 70.6 [44.0 to 89.7]

ADVERSE EVENTS:
Time Frame: up to 72 weeks
Groups:
- Vaniprevir 300 mg Bid + Peg-IFN + RBV: Participants received vaniprevir 300 mg twice daily in combination peg-IFN 180 mcg weekly and RBV 1000 or 1200 mg administered as a divided dose twice daily.
- Vaniprevir 600 mg Bid + Peg-IFN + RBV: Participants received vaniprevir 600 mg twice daily in combination peg-IFN 180 mcg weekly and RBV 1000 or 1200 mg administered as a divided dose twice daily.
Arm/Group | Vaniprevir 300 mg Bid + Peg-IFN + RBV | Vaniprevir 600 mg Bid + Peg-IFN + RBV
Serious Adverse Events (participants affected / at risk) | 4/21 | 1/24
Other Adverse Events (participants affected / at risk) | 21/21 | 23/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vaniprevir 300 mg Bid + Peg-IFN + RBV (N=21) | Vaniprevir 600 mg Bid + Peg-IFN + RBV (N=24)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vaniprevir 300 mg Bid + Peg-IFN + RBV (N=21) | Vaniprevir 600 mg Bid + Peg-IFN + RBV (N=24)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (3) | 2 (3)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (3) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 9 (14)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Flatulence (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 3 (3)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 3 (3)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 3 (3)
Nausea (Gastrointestinal disorders) | 8 (8) | 14 (17)
Vomiting (Gastrointestinal disorders) | 3 (4) | 2 (4)
Asthenia (General disorders) | 4 (4) | 6 (6)
Fatigue (General disorders) | 7 (7) | 5 (5)
Influenza like illness (General disorders) | 3 (4) | 4 (4)
Irritability (General disorders) | 2 (2) | 3 (3)
Pyrexia (General disorders) | 5 (6) | 3 (3)
Nasopharyngitis (Infections and infestations) | 2 (2) | 3 (4)
Urinary tract infection (Infections and infestations) | 3 (4) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 2 (7)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (3)
Weight decreased (Investigations) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (3) | 5 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (5)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Dizziness (Nervous system disorders) | 2 (4) | 3 (4)
Headache (Nervous system disorders) | 7 (7) | 9 (17)
Sciatica (Nervous system disorders) | 2 (2) | 0 (0)
Tremor (Nervous system disorders) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 5 (5)
Sleep disorder (Psychiatric disorders) | 3 (4) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 7 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5) | 6 (10)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission.